CLINICAL TRIAL: NCT01849679
Title: The Effect on Time After Extubation on Aspiration Risk
Brief Title: Post Extubation Dysphagia
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-0407
Record Dates: First submitted 2013-05-03; First posted 2013-05-08 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Severity of Aspiration in Post-extubated Subjects
Keywords: Dysphagia; extubation; aspiration
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Post-Extubation Subjects
  Interventions: Other: Evaluation of Swallowing

INTERVENTIONS:
Other: Evaluation of Swallowing — Evaluating for pharyngeal delay, pharyngeal stasis, and penetration/aspiration

SUMMARY:
The investigators hypothesize that aspiration will be more prevalent at two to four hours post-extubation but will resolve in the majority of patients by 24 to 26 hours post-extubation.

The purpose of the research is to investigate whether there is a difference in swallow function two to four hours after extubation (removal of breathing tube) compared to 24 hours after extubation. This information will help healthcare providers decide if it is necessary for people to wait 24 hours after extubation before they start eating and drinking.

ELIGIBILITY:
Inclusion Criteria:

* Patients that were intubated for more than 48 hours.
* Adults, 18 and over
* All races
* Males and females
* Approval to participate in the study by the treating physician

Exclusion Criteria:

* Patients with a history of oropharyngeal dysphagia.
* Patients with neurological disorders associated with dysphagia including dementia, Parkinson's disease, multiple sclerosis, stroke, and ALS.
* Patients with a history of head and neck cancer or laryngeal surgery.
* Patients that are not candidate for FEES because of facial fractures, nothing by mouth (NPO) status for other procedures, elevated bleeding risk (patients on therapeutically dosed anticoagulant infusion or injection, platelet count less than 50,000, INR greater than 2.0, partial thromboplastin time greater than 1.5 times normal), decreased level of arousal/alertness, significant agitation, or inability to tolerate room air or nasal cannula oxygen for duration of FEES.
* Patients who are extubated after 1400 or on weekends (Friday, Saturday, or Sunday).
* Non-English Speakers will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intubated inpatients 18 years and older at the University of Wisconsin Hospital Trauma and Life Support Center.
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2013-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Severity of Aspiration per Evaluation | post-extubation at 2-4 hours and possibly 24-26 hours.
  Flexible Endoscopic Evaluation of Swallow (FEES - a measure of swallowing which will allow for the diagnosis of swallowing) will be recorded at between 2 to 4 hour after extubation. If penetration/aspiration is noted during the evaluation between 2 to 4 hours post-extubation, then a second FEES evaluation will be completed between 24 to 26 hours post-extubation.

CONTACTS AND LOCATIONS:
Overall Officials: Stevie Marvin, MS, Principal Investigator — Univeristy of Wisconsin
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States